CLINICAL TRIAL: NCT03013777
Title: An Open-Label Pilot Trial of Cognitive Behavioral Therapy in Familial Dysautonomia
Brief Title: A Trial of Cognitive Behavioral Therapy in Familial Dysautonomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01823
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Dysthymia; Anxiety Disorders; Familial Dysautonomia; Paroxysmal Hypertension; Autosomal Recessive Disease
Keywords: Familial dysautonomia
MeSH Terms: conditions — Dysthymic Disorder; Anxiety Disorders; Dysautonomia, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive behavioral therapy (CBT) (Experimental): The patient would participate in eight forty-five minute sessions of CBT with a mental health therapist. Cognitive behavioral therapy (CBT), defined as a program of interventions that utilize education to teach relaxation, healthy coping skills, stress management, assertiveness training in order to help the individual identify and correct maladaptive beliefs in combination with education to help practice symptom reduction and improve quality of life and function.
  Interventions: Behavioral: 8-week CBT Program

INTERVENTIONS:
Behavioral: 8-week CBT Program

SUMMARY:
To determine the effect of cognitive behavioral therapy (CBT) in the severity of anxiety and depression in adult patients with familial dysautonomia. Patients will be enrolled in an 8-week CBT program. All CBT sessions will be done either in person at the NYU Dysautonomia Center or over the phone to help accommodate disability and potential physical limitations of our patient population.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT), defined as a program of interventions that utilize education to teach relaxation, healthy coping skills, stress management, assertiveness training in order to help the individual identify and correct maladaptive beliefs in combination with education to help practice symptom reduction and improve quality of life and function. Patients will participate in eight forty-five minute sessions of CBT with a mental health therapist in order to help treat generalized anxiety disorder, anxiety disorder due to another medical condition (familial dysautonomia), major depressive disorder, persistent depressive disorder (dysthymia), substance/medication- induced depressive disorder, depressive disorder due to another medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FD (genetically confirmed)
* DSM-V criteria of major depressive disorder OR anxiety disorder
* STAI score ≥ 25 OR a PHQ-9 depression scale score ≥ 5 or greater
* Willing and able to complete 8 CBT sessions
* Maintain constant psychoactive medication through out study and no concurrent talk therapy from another therapist.

Exclusion Criteria:

* Currently suicidal or having current suicidal ideations
* Currently under psychiatric treatment for depression or anxiety
* Have started any psychoactive medication within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) depression scale | 8 Weeks
  Short, but comprehensive scale that consists specifically to the criteria for diagnosis in the DSM-V. The PHQ-9 is effective and sensitive as an instrument in establishing tentative depressive disorder diagnoses while also assessing severity of depressive symptoms. The brevity and criterion validity of the scale make it an appropriate, dual purpose instrument for assessing the severity of depressive disorder within a clinical trial.
Rosenberg Self-Esteem Scale | 8 Weeks
  10-item questionnaire that objectively measures global self-worth. The Rosenberg Self-Esteem scale is a 10-item questionnaire that objectively measures global self-worth. The Rosenberg self-esteem scale is a 10-item scale scored using a four-point response. The scale has extensive and acceptable reliability and validity, both convergent and discriminant
State-Trait Anxiety Inventory (STAI) | 8 Weeks
  The STAI has 40 items, 20 items for each of the S-Anxiety and T-Anxiety sub scales. The STAI was chosen for brevity while also providing a broad coverage of DSM V diagnostic criteria for anxiety. The STAI has proven efficacy in measuring valid self-reports of anxiety symptoms and propensity for anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States